CLINICAL TRIAL: NCT05259371
Title: A 16-Week, Multi-Center, Open-Label, Exploratory Study to Evaluate the Safety and Efficacy of the Application of Pulse Electrical Stimulation Around the Eye in Early to Moderate Dry Age-Related Macular Degeneration
Brief Title: Study of Application of Transcutaneous Pulsed Electrical Stimulation Around Eye in Age-related Macular Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NE_RTN_002
Record Dates: First submitted 2022-02-11; First posted 2022-02-28 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Early to Moderate Dry Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; Macular degeneration; Early to Moderate Dry AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: • Experimental: Transcutaneous Pulsed Electrical Stimulation Treatment Patients wear our clinical trial device 30mins once a day for 16weeks. Device: Nu eyne M02
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous Pulsed Electrical Stimulation Treatment (Experimental): Patients wear our clinical trial device 30mins once a day for 16weeks. Device: Nu eyne M02
  Interventions: Drug: Transcutaneous Pulsed Electrical Stimulation (Device: Nu Eyne M02)

INTERVENTIONS:
Drug: Transcutaneous Pulsed Electrical Stimulation (Device: Nu Eyne M02) — Pulse Electrical Stimulation Patients wear our clinical trial device 30mins once a day for 16weeks.

SUMMARY:
This study aims to evaluate the safety and efficacy of applying pulse electrical stimulation around eyes of age-related macular patients.

DETAILED DESCRIPTION:
Duration of study period(per participant): Screening period(0-4weeks), Intervention period(16weeks) Patient needs to visit site at least 5 times(Screening, V2, V3, V4, V5). V2 can be done with screening visit. Visit 3, 4, 5 is 2weeks, 6weeks, and 16weeks after visit 2(Baseline).

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* Has a confirmed diagnosis of early to moderate AMD

  * According to Staging of age-related macular degeneration of Beckman Initiative for Macular Research Classification Committee

    * early AMD: Medium drusen(>63 μm; ≤125 μm) and No AMD pigmentary abnormalities
    * moderate AMD: Large drusen(>125 μm) and/or Any AMD pigmentary abnormalities
* Best Corrected Visual Acuity [BCVA] of 20/200 or better measured by Early Treatment Diabetic Retinopathy Study(ETDRS) Charts
* A person who voluntarily agreed to participate in this clinical trial

Exclusion Criteria:

* Subject who is observed to have a atrophy of 175 micrometers or more in diameter invading the fovea on fundus examination or fundus autofluorescent with more than one eye
* Subject who is observed to have exudative macular degeneration on fundus examination or optical coherence tomography(OCT) with more than one eye
* Has a history of intravitreal injection, laser treatment, etc.
* Has eye pathology other than early age-related macular degeneration that may affect the outcome of clinical trials.
* Has a history of vitrectomy due to macular disease or cataract surgery within 1 month
* Has a disease that is judged to be difficult to interpret an ophthalmic imaging examination due to ocular media opacity
* Has a history of uncontrollable systemic chronic disease(diabetes mellitus) or malignancy(cases that have not recurred for more than 5 years after complete recovery are excluded)
* Autoimmune disease(Sjögren's syndrome, Rheumatoid arthritis, systemic lupus erythematosus, Graves' disease, etc.)
* Has a severe hearing impairment
* A person who is sensitive to orbit nerve stimulation and cannot be treated.
* Has a history of substance and/or alcohol abuse
* Has a confirmed diagnosis of psychiatric disease(depression, schizophrenia, bipolar disorder, dementia, etc)
* Those who participated in other clinical trials within 30 days of the screening visit
* Those who are judged to have "other reasons for prohibition of use" of our clinical trial medical device: heart-related problems. seizure. Patients transplanted metal or electronic device in head & neck including deep brain stimulation device. Patient suffering from unknown pain. Patients with implantable or wearable cardioverter defibrillator. Patients who are warned not to use out clinical trial device or is prohibited from using it. (Dental implants are accepted.)
* In the case of subjects judged by the researcher that it would be difficult to participate in clinical trials
* Among female subjects who are likely to be pregnant, those who disagree to contraception in a medically permitted manner during this clinical trial period.

  * Medically permitted contraception: condom, Oral contraception that lasted for at least 3 months, contraceptive injection, contraceptive implant, intrauterine device, etc.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Safety Events | baseline ~ 16 weeks
  Check the safety issues(AE, SAE, etc.).

SECONDARY OUTCOMES:
Changes in contrast sensitivity | baseline, 6, 16 weeks
  Check the change of contrast sensitivity in the baseline, 6, 16 weeks
Changes in score of VFQ-25(National Eye Institute) | baseline, 6, 16 weeks
  Check the change of Changes in score of VFQ-25(National Eye Institute) in the baseline, 6, 16 weeks
Changes in best corrected visual acuity(Early Treatment Diabetic Retinopathy Study (ETDRS) Chart) | baseline, 6, 16 weeks
  Check the change of best corrected visual acuity in the baseline, 6, 16 weeks
Changes in drusen area using optical coherence tomography(OCT) | baseline, 6, 16 weeks
  Check the change of drusen area using optical coherence tomography(OCT) in the baseline, 6, 16 weeks
Changes in drusen volume using optical coherence tomography(OCT) | baseline, 6, 16 weeks
  Check the change of drusen volume using optical coherence tomography(OCT) in the baseline, 6, 16 weeks
Progression to advanced Age-related Macular Degeneration (AMD) using fundus autofluorescence(FAF) | baseline, 6, 16 weeks
  Check the Progression to advanced Age-related Macular Degeneration (AMD) using fundus autofluorescence(FAF) in the baseline, 6, 16 weeks
Progression to advanced Age-related Macular Degeneration (AMD) using fundus photography | baseline, 6, 16 weeks
  Check the Progression to advanced Age-related Macular Degeneration (AMD) using fundus photography in the baseline, 6, 16 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Nune Eye Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No